CLINICAL TRIAL: NCT06081309
Title: Electroencephalogram (EEG) Personalized Transcranial Magnetic Stimulation (eTMS) for Post-Traumatic Stress Disorder
Brief Title: EEG Personalized Transcranial Magnetic Stimulation (eTMS) for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eTMS-PTSD-001
Record Dates: First submitted 2023-10-01; First posted 2023-10-13 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Veterans; First Responders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is an open-label safety pilot study of EEG-based personalized TMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Open-Label active EEG-based personalized TMS treatment (Experimental): 20 sessions of EEG-based personalized TMS over a maximum of 21 days. Two sessions per treatment day. Each session consists of TMS treatment at 50% Motor Threshold, pulse frequency between 8-13 Hz. TMS delivery of 5 second pulse train, with an inter-train interval of 20 seconds. Session duration is 15 minutes. A rest period of at least 30 minutes is required between the 2 sessions in a treatment day.
  Interventions: Device: EEG-based personalized TMS

INTERVENTIONS:
Device: EEG-based personalized TMS — Transcranial Magnetic Stimulation (TMS), in which treatment is personalized based on the participant's Electroencephalogram (EEG)

SUMMARY:
This is an open-label safety pilot study of the Electroencephalogram (EEG) Transcranial Magnetic Stimulation (eTMS) treatment for Post-Traumatic Stress Disorder (PTSD). The recruitment goal is 30 participants who are United States Military veterans or first responders (e.g., firefighters, police, paramedics, etc.). The Study includes an EEG recording in order to determine the optimal treatment parameters for the eTMS system, followed by 10 in-office visits that take place over 21 total days. Two eTMS treatment sessions are administered during each office visit.

DETAILED DESCRIPTION:
eTMS-PTSD-001 is an open-label safety pilot study with a recruitment goal of 30 subjects, with 26 completers. The Study is intended to evaluate the safety aspects of eTMS in the target population. A maximum of 400 individuals will be screened in order to achieve the recruitment goal. The total number of days from the first participant enrolled to the last enrolled participant treated will be approximately 7 months.

Participants will be either Veterans or First Responders (e.g., emergency medical service provider, firefighter, or any other emergency response personnel), between 22-65 years of age. Participants may be male or female of any racial/ethnic background who meet the eligibility criteria. Participants will be recruited from the general public, and from veterans and first responder organizations.

The primary outcome for the Study will be the incidence, severity, relatedness, type, subsequent treatment/intervention required, and resolution status of adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent to participate in the study via signed Informed Consent
* Age 22 - 65 years
* Provisional diagnosis of PTSD
* Positive identification as either a Veteran, or First Responder (e.g., emergency medical service provider, firefighter, or any other emergency response personnel)

Exclusion Criteria:

* Uncontrolled medical, psychological or neurological condition
* Pregnant, or female unwilling to use effective birth control during the course of the trial
* Metal objects implanted in the head
* Past exposure to metal fragments or other metal sources in the head and neck
* Current participation in any interventional research protocol
* History of any type of Electroconvulsive Therapy (ECT) or TMS
* History of stroke or intracranial lesion, or increased intracranial pressure
* History or epilepsy or seizure
* Family history of epilepsy or seizure in 1st degree relative.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Phillips, PhD, Principal Investigator — Wave Neuroscience, Inc.
Locations (1):
- Wright State University, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers

REFERENCES:
- [Background] Bae EH, Schrader LM, Machii K, Alonso-Alonso M, Riviello JJ Jr, Pascual-Leone A, Rotenberg A. Safety and tolerability of repetitive transcranial magnetic stimulation in patients with epilepsy: a review of the literature. Epilepsy Behav. 2007 Jun;10(4):521-8. doi: 10.1016/j.yebeh.2007.03.004. Epub 2007 May 9. PMID 17493877
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Caulfield KA. Is accelerated, high-dose theta burst stimulation a panacea for treatment-resistant depression? J Neurophysiol. 2020 Jan 1;123(1):1-3. doi: 10.1152/jn.00537.2019. Epub 2019 Sep 25. PMID 31553674
- [Background] Corlier J, Carpenter LL, Wilson AC, Tirrell E, Gobin AP, Kavanaugh B, Leuchter AF. The relationship between individual alpha peak frequency and clinical outcome with repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder (MDD). Brain Stimul. 2019 Nov-Dec;12(6):1572-1578. doi: 10.1016/j.brs.2019.07.018. Epub 2019 Jul 25. PMID 31378603
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434
- [Background] George MS, Wassermann EM, Williams WA, Steppel J, Pascual-Leone A, Basser P, Hallett M, Post RM. Changes in mood and hormone levels after rapid-rate transcranial magnetic stimulation (rTMS) of the prefrontal cortex. J Neuropsychiatry Clin Neurosci. 1996 Spring;8(2):172-80. doi: 10.1176/jnp.8.2.172. PMID 9081553
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Hunter AM, Minzenberg MJ, Cook IA, Krantz DE, Levitt JG, Rotstein NM, Chawla SA, Leuchter AF. Concomitant medication use and clinical outcome of repetitive Transcranial Magnetic Stimulation (rTMS) treatment of Major Depressive Disorder. Brain Behav. 2019 May;9(5):e01275. doi: 10.1002/brb3.1275. Epub 2019 Apr 2. PMID 30941915
- [Background] Janicak PG, O'Reardon JP, Sampson SM, Husain MM, Lisanby SH, Rado JT, Heart KL, Demitrack MA. Transcranial magnetic stimulation in the treatment of major depressive disorder: a comprehensive summary of safety experience from acute exposure, extended exposure, and during reintroduction treatment. J Clin Psychiatry. 2008 Feb;69(2):222-32. doi: 10.4088/jcp.v69n0208. PMID 18232722
- [Background] Jin Y, Phillips B. A pilot study of the use of EEG-based synchronized Transcranial Magnetic Stimulation (sTMS) for treatment of Major Depression. BMC Psychiatry. 2014 Jan 18;14:13. doi: 10.1186/1471-244X-14-13. PMID 24438321
- [Background] Jin Y, Kemp AS, Huang Y, Thai TM, Liu Z, Xu W, He H, Potkin SG. Alpha EEG guided TMS in schizophrenia. Brain Stimul. 2012 Oct;5(4):560-8. doi: 10.1016/j.brs.2011.09.005. Epub 2011 Oct 6. PMID 22019083
- [Background] Leuchter AF, Cook IA, Jin Y, Phillips B. The relationship between brain oscillatory activity and therapeutic effectiveness of transcranial magnetic stimulation in the treatment of major depressive disorder. Front Hum Neurosci. 2013 Feb 26;7:37. doi: 10.3389/fnhum.2013.00037. eCollection 2013. PMID 23550274
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Loo C, Sachdev P, Elsayed H, McDarmont B, Mitchell P, Wilkinson M, Parker G, Gandevia S. Effects of a 2- to 4-week course of repetitive transcranial magnetic stimulation (rTMS) on neuropsychologic functioning, electroencephalogram, and auditory threshold in depressed patients. Biol Psychiatry. 2001 Apr 1;49(7):615-23. doi: 10.1016/s0006-3223(00)00996-3. PMID 11297719
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Carpenter LL, Conelea C, Tyrka AR, Welch ES, Greenberg BD, Price LH, Niedzwiecki M, Yip AG, Barnes J, Philip NS. 5 Hz Repetitive transcranial magnetic stimulation for posttraumatic stress disorder comorbid with major depressive disorder. J Affect Disord. 2018 Aug 1;235:414-420. doi: 10.1016/j.jad.2018.04.009. Epub 2018 Apr 5. PMID 29677606
- [Background] Roelofs CL, Krepel N, Corlier J, Carpenter LL, Fitzgerald PB, Daskalakis ZJ, Tendolkar I, Wilson A, Downar J, Bailey NW, Blumberger DM, Vila-Rodriguez F, Leuchter AF, Arns M. Individual alpha frequency proximity associated with repetitive transcranial magnetic stimulation outcome: An independent replication study from the ICON-DB consortium. Clin Neurophysiol. 2021 Feb;132(2):643-649. doi: 10.1016/j.clinph.2020.10.017. Epub 2020 Nov 10. PMID 33243617
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Sakkas P, Mihalopoulou P, Mourtzouhou P, Psarros C, Masdrakis V, Politis A, Christodoulou GN. Induction of mania by rTMS: report of two cases. Eur Psychiatry. 2003 Jun;18(4):196-8. doi: 10.1016/s0924-9338(03)00048-8. PMID 12814856
- [Background] Wobrock T, Guse B, Cordes J, Wolwer W, Winterer G, Gaebel W, Langguth B, Landgrebe M, Eichhammer P, Frank E, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Malchow B, Schneider-Axmann T, Falkai P, Hasan A. Left prefrontal high-frequency repetitive transcranial magnetic stimulation for the treatment of schizophrenia with predominant negative symptoms: a sham-controlled, randomized multicenter trial. Biol Psychiatry. 2015 Jun 1;77(11):979-88. doi: 10.1016/j.biopsych.2014.10.009. Epub 2014 Oct 23. PMID 25582269
- [Background] Yesavage JA, Fairchild JK, Mi Z, Biswas K, Davis-Karim A, Phibbs CS, Forman SD, Thase M, Williams LM, Etkin A, O'Hara R, Georgette G, Beale T, Huang GD, Noda A, George MS; VA Cooperative Studies Program Study Team. Effect of Repetitive Transcranial Magnetic Stimulation on Treatment-Resistant Major Depression in US Veterans: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Sep 1;75(9):884-893. doi: 10.1001/jamapsychiatry.2018.1483. PMID 29955803
- [Background] Ziemann U. TMS and drugs. Clin Neurophysiol. 2004 Aug;115(8):1717-29. doi: 10.1016/j.clinph.2004.03.006. PMID 15261850
- [Background] Ziemann U, Reis J, Schwenkreis P, Rosanova M, Strafella A, Badawy R, Muller-Dahlhaus F. TMS and drugs revisited 2014. Clin Neurophysiol. 2015 Oct;126(10):1847-68. doi: 10.1016/j.clinph.2014.08.028. Epub 2014 Dec 4. PMID 25534482
- See also: Study Information Page — http://etmsfda.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The eTMS-PTSD-001 study is divided into two stages: (Stage 1) An Open-Label safety pilot study; and (Stage 2) a randomized double-blind sham-controlled study. The current record (NCT06081309) covers only Stage 1. The study details and results for Stage 2 of the study will be reported in a separate record.
Period: Overall Study
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Education Level [Count of Participants; unit: Participants]
  Less than 9th Grade | 0
  9th - 12th Grade, No Diploma | 0
  High School Diploma or Equivalent | 0
  Some College, No Degree | 7
  Associate Degree | 9
  Bachelor's Degree | 9
  Graduate or Professional Degree | 5
Marital Status [Count of Participants; unit: Participants]
  Never Married | 3
  Separated | 0
  Married | 21
  Divorced | 5
  Widowed | 1
Military/First Responder [Number; unit: participants]
  Military - Reservist | 0
  Military - National Guard | 0
  Military - Retiree | 3
  Military - Veteran | 19
  1st Responder - Emergency Medical | 0
  1st Responder - Firefighter | 4
  1st Responder - Police | 6
  1st Responder - Search and Rescue | 0
  1st Responder - Crisis Counselor | 0

OUTCOME MEASURES:

1. Primary Outcome: Number, Severity, Relatedness, Type, Subsequent Treatment/Intervention Required, and Resolution Status of Adverse Events (AEs) During the Study.
Description: Number - Number of adverse events reported. Note that each participant may have had more than one adverse event (AE).
  Severity - Number of adverse events that were mild, moderate, or severe. Relatedness - Number of adverse events that were not related, suspected, or definitely related to treatment.
  Type - Number of adverse events that were or were not Serious Adverse Events (SAEs).
  Subsequent treatment/intervention required - Number of adverse events that did or did not require subsequent treatment/intervention.
  Number of participants reporting at least one AE
Time Frame: Baseline and Final Measure, between 10-21 Days
Population: Analyzed the total number of Adverse Events (AEs) that occurred in the study.
Measure: Number; unit: Number of AEs
Units Other Than Participants: AEs
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
Number analyzed (Participants) | 30
Number analyzed (AEs) | 31
Number of AEs
  Adverse Event Intensity - Mild | 26
  Adverse Event Intensity - Moderate | 3
  Adverse Event Intensity - Severe | 2
  Adverse Event Relationship to Treatment - Not Related | 17
  Adverse Event Relationship to Treatment - Suspected | 5
  Adverse Event Relationship to Treatment - Definitely Related | 9
  Serious Adverse Event | 0
  Not a Serious Adverse Event | 31
  Subsequent treatment/intervention required | 0
  No subsequent treatment/required | 31

2. Secondary Outcome: Improvement in PTSD Symptoms as Measured by Drop in Score on the PTSD Checklist for DSM-5 (PCL-5)
Description: The Post Traumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Ed. (DSM-5), commonly referred to as PCL-5, is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. It is used to monitor symptom change during and after treatment. Each item is scored from 0 to 5 as the participant's estimate of the severity of the symptom (0 = Not at all, 1=A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely). The final score range is between 0-80. A lower score is considered better than a higher score.
Time Frame: Baseline and Final Measure, between 10-21 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
Number analyzed (Participants) | 30
score on a scale
  Baseline Measure | 52.2 (8.9)
  Final Measure | 22.9 (14.0)
  Change between Baseline and Final Measure | 29.3 (13.1)

3. Post Hoc Outcome: Number of Participants With at Least One Adverse Event
Description: The number of participants who experienced at least one Adverse Event in the study
Time Frame: Baseline and Final Measure, between 10-21 Days
Population: Analyzed the total number of participants with at least one Adverse Event (AE) in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
Number analyzed (Participants) | 30
Participants | 14

ADVERSE EVENTS:
Time Frame: Baseline and Final Measure, between 10-21 Days. In addition, any adverse events that occurred after the Final Measure until Study completion were included.
Description: In the study, some participants experienced more than one Adverse Event. Therefore, in the table, the total number of Adverse Events listed is greater than the number of participants experiencing an Adverse Event.
Arm/Group | Open-Label Active EEG-based Personalized TMS Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 14/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Active EEG-based Personalized TMS Treatment (N=30)
Headache (General disorders) | 9 (9)
Mild Headache (General disorders) | 7 (7)
Sinus Headache (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Irritability (General disorders) | 2 (2)
Mild Head Cold (General disorders) | 2 (2)
Bruise (General disorders) | 1 (1)
Short-term Sadness (Nervous system disorders) | 1 (1)
Local Site Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open-label safety study. With no sham control, it is not possible to determine a statistically significant outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT06081309/Prot_SAP_000.pdf